CLINICAL TRIAL: NCT01744743
Title: Preconceptional Thyroid Screening and Childhood Nerocognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government); Shanghai Municipal Health Bureau (Other Government)
Responsible Party: Principal Investigator, Xiaotian Li, Vice president, Cheif of Obstetrics Department, Obstetrics and Gynecology Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12XD1401300
Record Dates: First submitted 2012-10-20; First posted 2012-12-07 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Hypothyroidism
Keywords: preconception; hypothyroidism; neurocognitive development
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- preconception (Active Comparator): Participants will be included according to their first outpatient visiting time. Women with TSH≥97.5%th and/or FT4≤2.5%th will accept levothyroxine 150ug daily and follow-up every 4 weeks. Medical records include: a)maternal thyroid function at enrollment; b) Levothyroxine: length, dose, drug adverse effects; c)Early trimester of pregnancy: Down's screening; d)2nd trimester of pregnancy: fetal echocardiography; e)Whole course of pregnancy: maternal complications, maternal blood pressure at each visit, fetal growth; f)Pregnancy outcome: type of delivery, length of labor, type and timing of analgesia/anesthesia, Apgar scores, postpartum hemorrhage, fetal complications; g)Offspring cognitive assessment at 0-3 years old
  Interventions: Procedure: levothyroxine
- early conception (Active Comparator): Participants will be included according to their first outpatient visiting time before 15+6 gestational week. Women with TSH≥97.5%th and/or FT4≤2.5%th will accept levothyroxine 150ug daily and follow-up every 4 weeks. Medical records include: a)maternal thyroid function at enrollment; b) Levothyroxine: length, dose, drug adverse effects; c)Early trimester of pregnancy: Down's screening; d)2nd trimester of pregnancy: fetal echocardiography; e)Whole course of pregnancy: maternal complications, maternal blood pressure at each visit, fetal growth; f)Pregnancy outcome: type of delivery, length of labor, type and timing of analgesia/anesthesia, Apgar scores, postpartum hemorrhage, fetal complications; g)Offspring cognitive assessment at 0-3 years old
  Interventions: Procedure: levothyroxine
- late conception (Placebo Comparator): Participants will be included according to their first outpatient visiting time after 16 gestational week. Women with TSH≥97.5%th and/or FT4≤2.5%th will accept levothyroxine 150ug daily and follow-up every 4 weeks. Medical records include: a)maternal thyroid function at enrollment; b) Levothyroxine: length, dose, drug adverse effects; c)Early trimester of pregnancy: Down's screening; d)2nd trimester of pregnancy: fetal echocardiography; e)Whole course of pregnancy: maternal complications, maternal blood pressure at each visit, fetal growth; f)Pregnancy outcome: type of delivery, length of labor, type and timing of analgesia/anesthesia, Apgar scores, postpartum hemorrhage, fetal complications; g)Offspring cognitive assessment at 0-3 years old
  Interventions: Procedure: levothyroxine

INTERVENTIONS:
Procedure: levothyroxine — Women with TSH≥97.5%th and/or FT4≤2.5%th will accept levothyroxine 150ug daily and follow-up every 4 weeks.

SUMMARY:
To assess the effect of universal preconception hypothyroidism for maternal pregnancy outcome, and 0-3yrs offspring neurocognitive ability and IQ score.

DETAILED DESCRIPTION:
Epidemic evidence and animal studies suggested that hypothyroidism is related with maternal pregnancy outcome, offspring cognitive ability. Negro's study found improved maternal health in those screened in early trimester; while Lazarus et al. reported no significant offspring IQ score at 3yrs in universal screening in early trimester. Currently, it lacks evidence of universal pre-conception screening for maternal pregnancy outcome and offspring cognitive development, motivation ability, attention. China Governmental Health Department has included thyroid function screening into preconception in 2011. The investigators hypothesize that pre-conception effective treatment may be helpful for decrease possible negative effects on maternal and offspring health, instead of early trimester.

ELIGIBILITY:
Inclusion Criteria:

1. Preconceptional group：TSH ≥ 97.5%th and/or FT4 ≤ 2.5%th
2. age: 18-55
3. those who can obey the rules of this study and assign the consent

Exclusion Criteria:

1. age: less than 18 or more than 55
2. multiple pregnancy
3. thyroid tumor disease history
4. those who cannot obey the rules of this study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Offspring neurocognitive assessment at 0-3 yrs | 3 months, 6 months, 1 year, 2 years, 3 years
  Peabody scale, Griffith scale
Offspring IQ assessment at 0-3 yrs | 3 months, 6 months, 1 year, 2 years, 3 years
  Wechsler Preschool Intelligence Scale at 1, 2, 3-year-old

SECONDARY OUTCOMES:
Incidence of neonatal hypothyroid and complications | up to 28 days of birth
  neonatal hypothyroid function, NICU rate, neonatal death rate

OTHER OUTCOMES:
Incidence of maternal complications | up to 42 days postpartumn
  preeclampsia, GDM, maternal death rate, maternal hemorrhage rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiaotian Li, MD, PhD, Principal Investigator — Obstetrics and Gynecology Hospital, Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhao Z, Zhou Q, Zhao H, Xiong Y, Li X. Association between levothyroxine treatment for maternal subclinical hypothyroidism with negative TPOAb and early child neurodevelopment: A prospective real-world clinical trial. Acta Obstet Gynecol Scand. 2023 Sep;102(9):1183-1192. doi: 10.1111/aogs.14602. Epub 2023 Jul 13. PMID 37443452
- [Derived] Zhou Q, Wang C, Xu H, Li X. Impact of Preconception Treatment Initiation for Hypothyroidism on Neurocognitive Function in Children. J Clin Endocrinol Metab. 2020 Nov 1;105(11):dgaa565. doi: 10.1210/clinem/dgaa565. PMID 32841335